CLINICAL TRIAL: NCT03903380
Title: Manual Therapy and Exercise With Mixed Reality With Hololens® Exercise Protocol in Chronic Neck Pain Subjects: Clinical Trial
Brief Title: Manual Therapy and Exercise With Mixed Reality With Hololens® Exercise Protocol in Chronic Neck Pain Patiens.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: problems recruiting the sample; derived from pandemic situation COVID-19
Sponsor: Centro Universitario La Salle (Other)
Collaborators: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Hector Beltran-Alacreu, Principal Investigator, Centro Universitario La Salle
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Holo-CNP
Record Dates: First submitted 2019-04-03; First posted 2019-04-04 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Neck Pain; Chronic Pain
Keywords: Virtual reality; Therapeuthic exercise; Quantitative sensory testing
MeSH Terms: conditions — Neck Pain; Chronic Pain | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MT treatment + Usual care exercise (Active Comparator): The intervention will be divided into two parts, the first one where MT treatment will take place and the second part where usual care exercise protocol will be introduced.
  The manual therapy protocol that will be used is the one proposed by Beltrán-Alacreu et al. (2015). The mentioned protocol consist of specific passive movements in the facet cervical joints, global mobilization of the cervical spine and high-velocity technique in the thoracic región.
  Interventions: Other: Manual Therapy and Usual care exercise protocol for neck pain
- MT treatment + Augmented reality (AR) exercises (Experimental): The intervention will be divided into two parts, the first one where MT treatment will take place and the second part where AR will be applied as an exercise method.
  The same manual therapy protocol will be used for both groups.
  For this group, the Microsoft HoloLens Development Edition device will be used, which is a holographic device that allows us to interact with high definition holograms in its environment. The application that will be used will be the Roboraid software, this app is a "shooter", which requires the cervical movement to move the pointer and be able to play.
  Interventions: Other: Manual Therapy and Augmented reality exercise protocol

INTERVENTIONS:
Other: Manual Therapy and Usual care exercise protocol for neck pain — Manual Therapy protocol between four to eight sessions and exercise protocol will be progressively added to the intervention (from the fouth session of MT approximately).
  Arms: MT treatment + Usual care exercise
Other: Manual Therapy and Augmented reality exercise protocol — Manual Therapy protocol between four to eight sessions and Augmented reality exercise protocol will be progressively added to the intervention (from the fouth session of MT approximately).
  Arms: MT treatment + Augmented reality (AR) exercises

SUMMARY:
Currently, cervical pain is the second most frequent musculoskeletal disorder, which generates an important impact on the function and quality of life. It is estimated that its anual prevalence for the general population can reach 50%.

Non-specific cervical pain attends without signs or symptoms of structural or neurological pathology, its etiology is unknown. However, it is related with joint and muscular structures. It has been observed a decrease in the strength and endurace of the deep cervical flexor muscles in 70% of patients with cervical pain; as well as motor control déficit and coordination alterations in the sinergy between the activity of the superficial and deep musculature.

Also, phycosocial factors, as for example: behaviors of fear-avoidance, catastrophism, hypervigilancy, psychosocial stress and negative adaptative neuroplastic changes, may have an importante role in chronic musculoskeletal pain.

In the last years, RV has been used in clinical rehabilitation, being a reliable and valid tool, which allows the patient distration to virtual world and they have offered results like: decreased pain and fear of movement and also improvements in motor performance and neuroplasticity processes.

The aim of this single-blinded randomized novel pilot study is to observe the effects generated in motor variables, when a protocol of manual therapy combined with augmented reality as a method of exercise in subjects with non-specific cervical pain is applied; in comparaison with a protocol of manual therapy combined with conventional cervical exercises.

Different variables will be measured at the beginning and at the end of intervention. Also, they will be measured one month after the intervention to observe the changes produced in short term. These variables are: pain, function, satisfaction, propioception, endurance, as well as phychological and somatosensory variables.

ELIGIBILITY:
Inclusion Criteria:

* - Men and women.
* Age: 18-65 years old.
* Persistent neck pain for at least 3 month or intermittent neck pain for 6 month or more.
* 5 points or 10% at the Neck Disability Index questionnaire.

Exclusion Criteria:

* Cervical whiplash (10 years before)
* Cervical fractures.
* Vestibular pathology.
* Epilepsy or other neurological condition.
* Systemic diseases.
* Cardiovascular or respiratory disorders that affect physical performance.
* Lasik eye surgery.
* Fibromyalgia
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Neck Disability Index (NDI) | change measures (Baseline, 4 weeks)
  A self-completed questionnaire based on Owestry Scale for low back pain. It is one of the most used questionnaires in the evaluation of cervical pain. Evaluates the disability level.
Cervical Joint Position Error Test: | change measures (Baseline, 4 weeks)
  This test is used to assess proprioception at the cervical level and the error in joint position sensation
Resistance test of the neck flexor muscles | change measures (Baseline, 4 weeks)
  To perform this test that will give us the resistance in seconds, the therapist lifts

SECONDARY OUTCOMES:
Tampa Scale for Kinesiophobia(TSK-11) | change measures (Baseline, 4 weeks)
  Self-report that assesses fear related to musculoskeletal pain. It is composed of 11 statements, in which the patient will have to rate from 1 to 4, being 1 totally in disagreement and 4 totally in agreement. The scores will range from 11 to 44 points, the higher the score the greater the fear of pain related to the movement.
Q Sense (Quantitative termal thresholds: cold and heat) | change measures (Baseline, 4 weeks)
  The thermotest Q-sense evaluates quantitatively the termal thresholds such as cold and heat, as well as the sensation of pain due to heat or cold. It provides an comprehensive somatosensory profile. It has been shown that in patients with sensory disorders of different etiologies, the sensory quantitative tests are considered as an useful/valuable diagnostic tool, which have good interobserver and test-retest reliability
Pain (VAS) | change measures (Baseline, 4 weeks)
  is a scale of 100 mm, in which the patient must make a mark to indicate the intensity of its pain, being the minimum value 0, which represents the absence of pain and the maximum value is 10, representing the worst pain.
Evaluation of User Satisfaction with Auxiliary Device Technology (QUEST 2.0) | change measures (Baseline, 4 weeks)
  This consists of 12 questions, each one of which the participant should circle with a circle the number that best describes his or her degree of satisfaction from 1 to 5 (1 being unsatisfied and 5 very satisfied)
System Usability Scale (SUS) | change measures (Baseline, 4 weeks)
  It consists of 10 questions and the participant should dial the number that best describes their degree of satisfaction from 1 to 5 (1 being unsatisfied and 5 very satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Josue Fernandez-Carnero, PhD, Study Chair — Universidad Rey Juan Carlos
Locations (1):
- IRF La Salle, Madrid, Madrid, Spain